CLINICAL TRIAL: NCT04592575
Title: Determining the Incidence of Vestibular Dysfunction in Traumatic Brain Injury Patients Admitted to Acute Inpatient Rehabilitation
Brief Title: Determining the Incidence of Vestibular Dysfunction in Traumatic Brain Injury Patients
Status: Completed | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, David Ripley, Principle Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00212535
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Brain Injuries, Traumatic
Keywords: Traumatic Brain Injury; Acute TBI; Vestibular Dysfunction
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI that are positive on screening tool: Patients that are identified on the AbilityLab Vestibular screening tool as possibly having vestibular dysfunction
  Interventions: Other: Vestibular Evaluation
- TBI patients not positive on screening tool: Patients that are not identified on the Ability Lab Vestibular screening tool as possibly having vestibular dysfunction
  Interventions: Other: Vestibular Evaluation

INTERVENTIONS:
Other: Vestibular Evaluation — Each patient will have a full vestibular evaluation by a physical therapist

SUMMARY:
The purpose of this study is to determine the incidence of vestibular dysfunction in traumatic brain injury patients admitted to acute inpatient rehabilitation. This study also seeks to validate the AbilityLab Vestibular Screening Tool (AVeST) and the AVeST+, tools designed to quickly screen individuals for vestibular dysfunction following traumatic brain injury.

DETAILED DESCRIPTION:
There are approximately 2.5 million hospital visits in the US each year for traumatic brain injury. Vestibular dysfunction is a common sequela of traumatic brain injury (TBI) affecting up to 50% of TBI patients at 5 years after injury. It is one of the most distressing problems for caregivers following TBI. Further complicating this issue is the fact that many individuals with TBI underestimate the severity of their balance deficits, which may further increase the risk of falls and subsequent injury. Sitting balance on admission to inpatient rehabilitation following TBI has been found to be one of the strongest predictors of functional status at discharge from inpatient rehabilitation. Due to the multifaceted presentation of vestibular dysfunction, evaluation is challenging, and there is currently no standardized approach to screening. While the incidence of vestibular dysfunction has been studied in mild TBI (mTBI) and sports related concussions, there is a gap in the literature regarding the incidence of vestibular dysfunction in moderate to severe TBI patients in acute inpatient rehabilitation.

The benefits of having an established vestibular dysfunction screening and rehabilitation program are multifold. Vestibular rehabilitation following TBI has demonstrated improvements in cognitive function, ability to return to activities of daily living, ability to return to work, and the need for assistance. While one prior single blind randomized controlled trial aimed to evaluate the effectiveness of a structured vestibular rehabilitation program in TBI individuals, there is a need for a large-scale study to evaluate the effectiveness of screening for vestibular dysfunction in order to create a systematic approach. Many TBI patients are not diagnosed with vestibular dysfunction until much later in their hospital course which impedes participation in therapy and likely has a detrimental effect on their rate of recovery. Identifying these patients earlier in their rehabilitation course will allow interventions that will improve and accelerate patient outcomes. An additional benefit of this study is to determine the incidence of vestibular dysfunction in moderate to severe TBI patients to outline the necessary resources to care for patients with this problem. Data collected will be utilized to validate the AVeST and the AVeST+. Additionally, this study will fill a gap in the literature in delineating the incidence of vestibular impairment in individuals with moderate to severe brain injury, a population heretofore not previously studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to an inpatient brain injury service at the Shirley Ryan Ability Lab with a history of moderate to severe traumatic brain injury, defined by an initial Glasgow coma scale (GCS) <13 and/or evidence of intracranial injury on neuroimaging
2. Able to complete vestibular screening evaluation
3. Age >18
4. Fluent in English

Exclusion Criteria:

1. Those with mild traumatic brain injury, defined by an initial Glasgow coma scale (GCS) >13
2. Those who are unable to reliably participate in and complete vestibular screening evaluation
3. Age <18
4. Individuals who do not speak English
5. Prior history of vestibular dysfunction

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic brain injury patients admitted to an inpatient rehabilitation facility
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
AbilityLab Vestibular Screening Tool (AVEST) | within the first few days of admission to acute inpatient rehabilitation
  a subjective questionnaire (yes/no questions) completed by a physician or therapist
AbilityLab Vestibular Screening Tool + (AVEST+) | within the first few days of admission to acute inpatient rehabilitation
  Physical examination and screen rated as impaired or not impaired

SECONDARY OUTCOMES:
Vestibular Evaluation by Physical Therapist | After screening tool completed and referral by physician to vestibular therapist
  Full oculomotor and vestibular exam to determine vestibular dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Holly Paczan, PT, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No